CLINICAL TRIAL: NCT03360045
Title: The Evaluation of Effectiveness of Nasal Compression With Tranexamic Acid Compared to Simple Nasal Compression and Merocel Packing
Brief Title: Comparing Effectiveness of Merocel and Packing With Tranexamic Acid in the Management of Anterior Epistaxis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Şeref Kerem Çorbacıoğlu, Associated professor, Kecioren Education and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71146310-511.06-E.223856
Record Dates: First submitted 2017-11-19; First posted 2017-12-02 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Tranexamic Acid; Epistaxis; Nasal Packing
MeSH Terms: conditions — Epistaxis | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Tranexamic acid group (Active Comparator): 500mg tranexamic acid is sprayed in the nose by atomizer spray, and then is applied nasal compression by manually.
  Interventions: Drug: Tranexamic Acid
- Placebo group (Placebo Comparator): 5ml normal saline is sprayed in the nose by atomizer spray, and then is applied nasal compression by manually.
  Interventions: Drug: Normal saline
- Merocel Group (Active Comparator): Merocel packing is applied.
  Interventions: Device: Merocel

INTERVENTIONS:
Drug: Tranexamic Acid — 500mg tranexamic acid is sprayed in the nose by atomizer spray, and then is applied nasal compression by manually.
  Arms: Tranexamic acid group
Drug: Normal saline — 5 cc normal saline is sprayed in the nose by atomizer spray, and then is applied nasal compression by manually.
  Arms: Placebo group
Device: Merocel — Merocel packing is applied.
  Arms: Merocel Group

SUMMARY:
Aim of this study is evaluate whether superior nasal compression with tranexamic acid to simple nasal compression and Merocel packing.

In this study, patients who presented with non-traumatic anterior epistaxis to emergency departments will be included in this study. Three different therapy option are created; first, nasal compression with tranexamic acid, second, simple nasal compression without any drugs. And third, packing with Merocel.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior epistaxis older than 18 year and accept to participate in the study

Exclusion Criteria:

* Patients younger than 18 years
* Patients who used anticoagulation therapy
* Patients who have hemodynamically instability
* Traumatic epistaxis
* Patients who have known bleeding disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Success rate of interventions to stop bleeding | First 15 minutes
  Percentages of numbers of patients who have stopped bleeding within first 15 minutes after nasal compression or Merocel packing
Numbers of patients who needs rescue treatment | After 15 minutes first intervention method.
  In patients who have unstoppable epistaxis within 15 minutes, Merocel packing will be applied as a rescue treatment. Numbers of these patients will be recorded.

SECONDARY OUTCOMES:
Re-bleeding | 24 hour
  Frequency of re-bleeding within first 24 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Keçiören Training and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Akkan S, Corbacioglu SK, Aytar H, Emektar E, Dagar S, Cevik Y. Evaluating Effectiveness of Nasal Compression With Tranexamic Acid Compared With Simple Nasal Compression and Merocel Packing: A Randomized Controlled Trial. Ann Emerg Med. 2019 Jul;74(1):72-78. doi: 10.1016/j.annemergmed.2019.03.030. Epub 2019 May 9. PMID 31080025